CLINICAL TRIAL: NCT03662321
Title: Prevalence and Vulnerability Factors of Active Cybersexuality Among Teenagers (15 - 17 Olds) in West Normandy.
Brief Title: Quantitative Study of Prevalence and Vulnerability Factors of Active Cyber Sexuality Among Teenagers in West Normandy
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-192
Record Dates: First submitted 2018-07-04; First posted 2018-09-07 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2018-02

CONDITIONS: Teenager; Sex Behavior
Keywords: teenager; sexuality; internet
MeSH Terms: conditions — Sexual Behavior; Sexuality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sexual behavior on the internet: this group of teenagers use internet for sexuality
- not sexual behavior on the internet: this group of teenagers doesn't use internet for sexuality

SUMMARY:
This study evaluates prevalence of active cybersexuality among teenagers (15-17 old) in West Normandy and find different factors of vulnerability that could induce this behaviour. Selection of teenagers in different schools (general, professional, agricultural, reintegration structure).

DETAILED DESCRIPTION:
the teen completes a questionnaire at the beginning of sexual education session. This questionnaire put in an anonymous box. After, there is a debate on the subject with the speaker, teenager ask questions about sexuality.

ELIGIBILITY:
Inclusion Criteria:

* all of teenagers participate a sexual education session

Exclusion Criteria:

* <15 old and 18 old and more
* the school doesn't want to participate
* one parent refuses that his adolescent participate. If requested exclusion, the group to which belongs the child is excluded
* teenager refuses to participate

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: population of teenagers of different school structures . make differences between the urban schools and the rural schools
Sampling Method: Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
prevalence of active cybersexuality | 20 minutes
  if teenagers send, receive or forward pictures or videos nude, use dedipix, participate to skin party, speak on chats. Evaluation by anonymous questionnaire distributed at the beginning of the session. They answered "yes" or "no" or "I don't want to answer" . If They answered "yes" to one question they were considered to be practicing cybersexuality

SECONDARY OUTCOMES:
factors of vulnerability that induce sexuality on the internet | 20 minutes
  factors of vulnerability are: gender, welfare, emotional bond with parents, accessibility of internet, use internet and social network, see pornography, addictive behavior, trauma in the past. Evaluation by anonymous questionnaire. Inside, Using an analog scale for the consumption of the internet and phone, more the number is important (the max was 10 hours and 200 sms) more the teenagers surfed in the internet. For the others questions , four answers are possible "yes very well", "yes, well", "not really" "not at all" more they answered not at all more it was a factor of vulnerability

CONTACTS AND LOCATIONS:
Overall Officials: CHU Caen, Principal Investigator — university hospital center
Locations (14):
- France (14):
  - Lycée de navarre, Alençon
  - Cfai Uimm, Caen
  - CIFAC, Caen
  - EPEI, Caen
  - ICEP CFA, Caen
  - Lycée Allende, Caen
  - Lycée Laplace, Caen
  - Lycée Millet, Cherbourg
  - La roquelle, Coutances
  - IME, Démouville
  - Lycée jules verne, Mondeville
  - MFR TRUN, Trun
  - MFR, Vimoutiers
  - Lycée marie curie, Vire

REFERENCES:
- [Background] Braun-Courville DK, Rojas M. Exposure to sexually explicit Web sites and adolescent sexual attitudes and behaviors. J Adolesc Health. 2009 Aug;45(2):156-62. doi: 10.1016/j.jadohealth.2008.12.004. Epub 2009 Feb 20. PMID 19628142
- [Background] Strassberg DS, McKinnon RK, Sustaita MA, Rullo J. Sexting by high school students: an exploratory and descriptive study. Arch Sex Behav. 2013 Jan;42(1):15-21. doi: 10.1007/s10508-012-9969-8. Epub 2012 Jun 7. PMID 22674035
- [Background] Temple JR, Paul JA, van den Berg P, Le VD, McElhany A, Temple BW. Teen sexting and its association with sexual behaviors. Arch Pediatr Adolesc Med. 2012 Sep;166(9):828-33. doi: 10.1001/archpediatrics.2012.835. PMID 22751805
- [Background] Strassberg DS, Cann D, Velarde V. Sexting by High School Students. Arch Sex Behav. 2017 Aug;46(6):1667-1672. doi: 10.1007/s10508-016-0926-9. Epub 2017 Jan 3. PMID 28050742
- [Background] Rice E, Gibbs J, Winetrobe H, Rhoades H, Plant A, Montoya J, Kordic T. Sexting and sexual behavior among middle school students. Pediatrics. 2014 Jul;134(1):e21-8. doi: 10.1542/peds.2013-2991. PMID 24982103